CLINICAL TRIAL: NCT04591756
Title: Effectiveness of Respiratory Protection During Simulated Resuscitation: a Prospective Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Andrew Barros, Assistant Professor, Department of Medicine, Pulmonary and Critical Care, University of Virginia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSR200209
Record Dates: First submitted 2020-10-12; First posted 2020-10-19 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Occupational Exposure
Keywords: Respirator; Cardiopulmonary resusitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N95 Filtering Facepiece Respirator (Active Comparator): Subjects will wear the model of filtering facepiece respirator that they are currently approved to wear
  Interventions: Other: Qualitative Fit Testing
- Elastomeric Half-Mask Respirator with P100 filters (Active Comparator): Subjects will wear the model of elastomeric half mask respirator that they are currently approved to wear.
  Interventions: Other: Qualitative Fit Testing

INTERVENTIONS:
Other: Qualitative Fit Testing — Qualitative fit testing with denatonium benzoate

SUMMARY:
The study hypothesizes that EHMRs with P100 filters will provide superior respiratory protection during simulated CPR compared to disposable N95 FFRs as measured by qualitative fit testing.

To this end, the study is a prospective observational cohort to evaluate the effectiveness of disposable FFRs and EHMR during simulated CPR. The primary endpoint will be subject report of detection of the testing agent during a 2 minute session of simulated chest compressions on a mannequin while wearing the respiratory protection that subjects routinely wear during the course of employment.

ELIGIBILITY:
Inclusion Criteria:

* Current use of respirator within last 7 days
* Completed fit test with respirator within last 2 years

Exclusion Criteria:

* Previous adverse reaction to fit testing or testing agent
* Development of any health problem that precludes use of a respirator since last occupational health evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Subject Detection of Testing Agent | 2 minutes
  Subject reported detection of testing agent

SECONDARY OUTCOMES:
Time to detection of testing agent | 2 minutes
  Time to subject reported detection of testing agent

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Barros, MD, Principal Investigator — University of Virginia
Locations (1):
- UVAHealth, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No